

## **Consent and Authorization Document**

Huntsman Intermountain Adolescent Young Adult and Cancer Health Insurance Tools

#### SUMMARY

The purpose of this Huntsman Intermountain Adolescent Young Adult (HIAYA) and Cancer Health insurAnce Tools (CHAT) study is to assess health insurance knowledge, barriers to becoming insured, and concerns about cost of care among adolescents and young adults (AYAs) with cancer.

We are doing this study because AYAs are more likely to be underinsured and have less experience health insurance than older patients. This study will compare two methods of educating participants about health insurance. Whether or not you take part in this study is entirely up to you. You are free to say yes or no. If you agree to participate in this study, you will be randomly (like the flip of a coin) put into to one of two groups.

As a participant in this study, you will be asked to complete two surveys, possibly participate in 4 videoconference sessions that discuss health insurance and then be interviewed about how well this program is working. This study team would be in contact with you for about 5 months. To thank you for your time and effort in this study, we will provide you with two \$20 gift cards, one after each survey.

There are some minimal risks for participating in this study include possible breach of confidentiality, or discomfort from answering study questions. There are no expected benefits for participating in this study, but you may learn more about health insurance.

## **STUDY PROCEDURES**

If you decide to join this study, you will be randomly assigned to **Group A** or **Group B**. You will be asked to take part in the study for about 5 months, which will span the study activities of the initial survey, the completion of the program, and a post-program survey. You may also be asked to complete an interview after these activities have been completed with a member of the study team.

Both Group A participants and Group B participants will participate in surveys.

- The surveys will be given at two different times at study enrollment and again about 2 months after that for a follow-up.
- We will ask you to answer a set of questions about your medical history, basic demographic information, and your insurance experiences, knowledge, and coverage history.
- Answering these questions should take no more than approximately 15 minutes each time. You do not have to answer any questions that make you uncomfortable.



University of Utah Institutional Review Board Exemption 3/2/2020 If you are assigned to **Group A**, the following things will happen:

- Insurance Education Sessions (videoconferencing-based options available): The study team will arrange 4 health insurance educational sessions between you and a patient navigator that will occur every other week over 2 months. The sessions will be 30 minutes long and can be delivered to you inperson, over the phone or through an online videoconference portal. If needed, this will allow you to take part in the sessions on a device of your choosing (smartphone, tablet, laptop, desktop computer, etc.) You may opt out of the sessions at any time.
- <u>Mailing of a Health Insurance Information Booklet:</u> The study will also send you a mailed copy of "The Healthcare Law: How it Can Help People with Cancer and Their Families", a booklet developed by the American Cancer Society.
- <u>Exit Interview (videoconferencing-based options available):</u> The study will contact you to schedule an interview upon your completion of the health insurance education sessions. This one time interview will be conducted by a study team member, and will be occur in-person, over the phone or through an online videoconference portal. If needed, this will allow you to take part in the sessions on a device of your choosing (smartphone, tablet, laptop, desktop computer, etc.) Interviews are estimated to be about 20 minutes long.

If you are assigned to **Group B**, the following things will happen:

- You will be able utilize the standard patient navigation services as usual.
- Mailing of a Health Insurance Information Booklet: The study will send you a mailed copy of "The Healthcare Law: How it Can Help People with Cancer and Their Families", a booklet developed by the American Cancer Society.

## **PERSON TO CONTACT**

<u>Study Team</u>: If you have any questions, complaints, or if you feel you have been harmed by this research please contact Dr. Anne Kirchhoff at the University of Utah by email at <u>anne.kirchhoff@hci.utah.edu</u> or via phone at 801-587-4084, Monday-Friday 9 a.m. to 4 p.m.

<u>Institutional Review Board</u>: Contact the Institutional Review Board (IRB) if you have questions regarding your rights as a research participant. Also, contact the IRB if you have questions, complaints or concerns which you do not feel you can discuss with the investigator. The University of Utah IRB may be reached by phone at (801) 581-3655 or by e-mail at <u>irb@hsc.utah.edu</u>.

<u>Research Participant Advocate</u>: You may also contact the Research Participant Advocate (RPA) by phone at (801) 581-3803 or by email at <u>participant.advocate@hsc.utah.edu</u>.



#### **VOLUNTARY PARTICIPATION**

Research studies include only people who choose to take part. You can tell us that you don't want to be in this study. You can start the study and then choose to stop the study later. This will not affect your relationship with the investigator or anyone on your healthcare team.

#### **COSTS AND COMPENSATION TO PARTICIPANTS**

There are no costs to being in this study. You may be compensated by completing surveys, completing exit interview. In total you will receive between \$40 and \$60 in gift cards for full participation.

## **RISKS**

There are some small risks related to taking part in this study. Questions and discussion about health insurance can be psychologically stressful. As a reminder, you may choose not to answer or discuss any questions that you do not want to and may decide to drop out of the study at any time. There is also a small risk of loss of confidentiality, but we do everything possible to keep your information secure.

#### **BENEFITS**

There are no direct benefits for taking part in this study. You may learn information about health insurance coverage and access. However, we hope the information we get from this study may help develop a greater insight of AYA cancer patients and insurance understanding in the future.

#### **AUTHORIZATION FOR USE OF YOUR PROTECTED HEALTH INFORMATION**

Signing this document means you allow us, the researchers in this study, and others working with us to use some information about your health for this research study.

This is the information we will use and include in our research records:

- Demographic and identifying information like name, current age, gender, insurance information, address, telephone number, and email address.
- Related medical information about you like personal and family medical history, primary diagnosis, age at diagnosis, current and past medications or therapies.

## How we will protect and share your information:

- We will do everything we can to keep your information private but we cannot guarantee this. Study information will be kept in a secured manner and electronic records will be password protected. Study information may be stored with other information in your medical record. Other doctors, nurses, and third parties (like insurance companies) may be able to see this information as part of the regular treatment, payment, and health care operations of the hospital. We may also need to disclose information if required by law.
- In order to conduct this study and make sure it is conducted as described in this form, the research records may be used and reviewed by others who are working with us on this research:



University of Utah Institutional Review Board Exemption 3/2/2020

- Members of the research team at University of Utah, Huntsman Cancer Institute, Intermountain Health Care
- The University of Utah Institutional Review Board (IRB), who reviews research involving people to make sure the study protects your rights;
- If we share your information with groups outside of University of Utah Health or Intermountain Healthcare we will not share your name or identifying information. We will label your information with a code number, so they will not know your identity.
- If you do not want us to use information about your health, you should not be part of this research. If you choose not to participate, you can still receive health care services at University of Utah Health and Intermountain Healthcare.

## What if I decide to Not Participate after I sign the Consent and Authorization Form?

You can tell us anytime that you do not want to be in this study and do not want us to use your health information. You can also tell us in writing. If you change your mind, we will not be able to collect new information about you, and you will be withdrawn from the research study. However, we can continue to use information we have already started to use in our research, as needed to maintain the integrity of the research.

This authorization does not have an expiration date.

# **CONSENT**

I confirm that I have read this consent and authorization document and have had the opportunity to ask questions. I will be given a signed copy of the consent and authorization form to keep.

I agree to participate in this research study and authorize you to use and disclose health information about me for this study, as you have explained in this document.

| Participant's Name | |
|---------------------------------------------------------|----------|
| Participant's Signature | <br>Date |
| raiticipant's Signature | Date |
| Name of Person Obtaining Authorization and Consent | |
| Signature of Person Obtaining Authorization and Consent | Date |

